CLINICAL TRIAL: NCT03031327
Title: A 2 Weeks, Randomized, Double-masked, Controlled Study to Assess Tolerability, Safety, Permanence on the Ocular Surface, Efficacy of Lubricin (20 and 50 μg/ml) vs Sodium Hyaluronate 0.18% in Ocular Discomfort Following Refractive Surgery.
Brief Title: Safety and Efficacy of 2 Concentrations of Lubricin vs Sodium Hyaluronate in Ocular Discomfort After Refractive Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUB0116MD; CIV-15-05-013553 (Other: EudaMed)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Ocular Discomfort
Keywords: Ocular Discomfort Following Refractive Surgery; Refractive Surgery; sodium hyaluronate; HA; Vismed®; Lubricin
MeSH Terms: conditions — Jacobs syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The packaging used for the comparator in the present investigation aimed at ensuring a complete masking of the test IMD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lubricin 20µg/ml (Experimental): Lubricin 20µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Interventions: Device: Lubricin 20µg/ml
- Lubricin 50µg/ml (Experimental): Lubricin 50µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Interventions: Device: Lubricin 50µg/ml
- Sodium hyaluronate (Active Comparator): Vismed® 0.18% Sodium hyaluronate (HA) eye drops
  Comparator was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Interventions: Device: Sodium hyaluronate 0.18%

INTERVENTIONS:
Device: Lubricin 20µg/ml — Lubricin 20µg/ml eye drops
  Arms: Lubricin 20µg/ml
Device: Lubricin 50µg/ml — Lubricin 50µg/ml eye drops
  Arms: Lubricin 50µg/ml
Device: Sodium hyaluronate 0.18% — Sodium hyaluronate (HA) 0.18% eye drops
  Other Names: Vismed®
  Arms: Sodium hyaluronate

SUMMARY:
The objective of this study was to evaluate tolerability, safety, permanence on the ocular surface and efficacy of Lubricin (20 and 50 μg/mL) eye drops vs Sodium Hyaluronate (Vismed®) 0.18% eye drops in patients with ocular discomfort following refractive surgery.

Primary objectives:

* Tolerability using a Visual analogue scale (VAS) for dryness, foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia;
* Treatment-emergent adverse events (TEAEs), assessed throughout the study.

Secondary objectives:

* Ocular surface vital staining with Fluorescein (Oxford scale)
* Schirmer-I test (without anaesthesia);
* Permanence of Lubricin on the Ocular Surface Tear film break-up time (TFBUT);
* Best corrected distance visual acuity (BCDVA);
* SANDE questionnaire scores - discomfort improvement entity;
* SANDE questionnaire scores - discomfort improvement speed;
* Signs evaluated by Slit lamp examination (SLE) (blepharitis, eyelid hyperemia/oedema, lashes, conjunctiva hyperemia);
* Intraocular pressure (IOP) ;
* Corneal sensitivity by Cochet-Bonnet aesthesiometry.

All parameters were evaluated at V1 (Day 1 - Baseline), V2 (Day 15±2) and V3 (Day 22±2/ETV).

DETAILED DESCRIPTION:
This study was a 2 week randomized (1:1:1), controlled, double-masked, parallel group, pre-market study to evaluate tolerability, safety, permanence on the ocular surface and efficacy of Lubricin (20 and 50 μg/mL) eye drops vs Sodium Hyaluronate (Vismed®) 0.18% eye drops in patients with ocular discomfort following refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older;
2. Patients undergone ocular refractive surgery within 6 months from V1 - Day 1;
3. Patients with ocular discomfort defined as SANDE score ≥ 30 at baseline;
4. Average VAS score (dryness, foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia) ≥ 25 mm;
5. Best corrected distance visual acuity (BCDVA) score ≥ 0.1 decimal units in both eyes at the time of study enrolment;
6. Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the Ethics Committee for the current study.

Exclusion Criteria:

1. Patients with a severe Dry Eye condition (severity level 4 according to the Report of the International Dry Eye Workshop -DEWS, 2007);
2. Best corrected distance visual acuity (BCDVA) score of < 0.1 decimal units in either eye at the time of study enrolment;
3. Evidence of an active ocular infection in either eye;
4. History or presence of ocular surface disorders other than ocular discomfort in either eye;
5. Use of any ocular topical medication other than the study medications for the treatment of ocular diseases including artificial tears during the study period;
6. Use of topical cyclosporine, topical corticosteroids or any other topical medication for the treatment of dry eye in either eye within 30 days of study enrolment;
7. History of any ocular surgery (excluding laser or refractive surgical procedures) in either eye within 30 days before study enrolment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period;
8. Known hypersensitivity to one of the components of the study or procedural medications;
9. Participation in another clinical study at the same time as the present study or within 90 days of screening/baseline visit;
10. History of drug, medication or alcohol abuse or addiction;
11. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

    1. are currently pregnant or,
    2. have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
    3. intend to become pregnant during the study treatment period or,
    4. are breast-feeding or,
    5. not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or IUD (intrauterine device ) during the entire course of and 30 days after the study treatment periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD-PhD, Study Director — Dompé Farmaceutici S.p.A
Locations (1):
- Dipartimento "Organi di senso" Università La Sapienza- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty (30) patients (10 per arm) randomized 1:1:1 to Lubricin 20 μg/mL eye drops solution or Lubricin 50 μg/mL eye drops solution or sodium hyaluronate (HA) 0.18% eye drops solution were enrolled, randomised and treated. The enrolled and safety analysis sets included all 30 enrolled and treated subjects, while the full analysis set (FAS) included 29 subjects and excluded one of the 2 discontinued subjects due to major protocol deviations.
Groups:
- Lubricin 20µg/ml: Lubricin 20µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 20µg/ml: Lubricin 20µg/ml eye drops
- Lubricin 50µg/ml: Lubricin 50µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 50µg/ml: Lubricin 50µg/ml eye drops
- Sodium Hyaluronate: Vismed® 0.18% Sodium hyaluronate (HA) eye drops
  Comparator was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Sodium hyaluronate 0.18%: Sodium hyaluronate (HA) 0.18% eye drops
Period: Overall Study
Arm/Group | Lubricin 20µg/ml | Lubricin 50µg/ml | Sodium Hyaluronate
Started | 10 | 10 | 10
Full Analysis Set Population (FAS) | 10 | 10 | 9
Safety Population (SAF) | 10 | 10 | 10
Patients in Which Left Eye is the Study Eye | 6 | 6 | 5
Patients in Which Right Eye is the Study Eye | 4 | 4 | 5
Completed | 10 | 9 | 9
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographics are based on the Enrolled set (n=30)
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubricin 20µg/ml | Lubricin 50µg/ml | Sodium Hyaluronate | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 10 | 29
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (14.4) | 37.4 (12.2) | 39.1 (9.7) | 38.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 17
  Male | 4 | 4 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline (Day 1 Pre-dose) in Ocular Tolerability Using a Visual Analogue Scale (VAS)
Description: A global ocular tolerability score was determined using a 100 mm Visual Analogue Scale (VAS) on which 0 meant no symptoms and 100 meant the worst possible discomfort. This evaluation was to be performed before any ophtalmic assessment at each scheduled visit. Specific ocular symptoms measured with the VAS included: foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia. The patients evaluated their symptoms using the VAS giving the value they were feeling from none to an extreme value. The VAS scale was a straight horizontal line of fixed length (100 mm). The ends were defined as extreme limits of the parameter.
Time Frame: Day 1 (baseline = Visit 1) at pre-dose, 15, 30 min post-dose; Day 15±2 (= Visit 2) at pre-dose, 15, 30 min post-dose; Day 22±2 (= Visit 3)
Population: The Full Analysis Set (FAS) population included all randomised patients, who received and used at least once the investigational device (Lubricin or Vismed®). This analysis set was used for the efficacy analysis. Please note that for participants, study eye and non-study eye values were assessed and reported.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Groups:
- Lubricin 20µg/ml (FAS): Lubricin 20µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 20µg/ml: Lubricin 20µg/ml eye drops
- Lubricin 50µg/ml (FAS): Lubricin 50µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 50µg/ml: Lubricin 50µg/ml eye drops
- Sodium Hyaluronate (FAS): Vismed® 0.18% Sodium hyaluronate (HA) eye drops
  Comparator was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Sodium hyaluronate 0.18%: Sodium hyaluronate (HA) 0.18% eye drops
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
mm
  Dryness - Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 1 (15 min) | -22.8 (13.2) | -30.1 (15.4) | -20.9 (14.2)
  Dryness - Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 1 (30 min) | -20.9 (13.3) | -29.3 (18.6) | -19.6 (11.9)
  Dryness - Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 15±2 (pre-dose) | -17.6 (17.0) | -17.3 (20.0) | -14.2 (12.2)
  Dryness - Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 15±2 (15 min) | -25.9 (15.4) | -33.3 (25.7) | -22.7 (10.6)
  Dryness - Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 15±2 (30 min) | -22.5 (15.1) | -29.8 (25.0) | -19.7 (10.8)
  Dryness - Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Dryness - Study eye - Day 22±2 | -5.9 (12.4) | -8.1 (6.4) | -4.4 (9.6)
  Dryness - Non Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 1 (15 min) | -18.7 (12.4) | -23.3 (18.4) | -22.7 (10.1)
  Dryness - Non Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 1 (30 min) | -18.4 (12.9) | -23.6 (20.8) | -19.7 (10.4)
  Dryness - Non Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 15±2 (pre-dose) | -10.8 (15.7) | -12.0 (19.1) | -10.2 (12.3)
  Dryness - Non Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 15±2 (15 min) | -19.5 (15.0) | -25.3 (25.2) | -22.2 (12.1)
  Dryness - Non Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 15±2 (30 min) | -17.2 (15.7) | -23.1 (25.3) | -17.8 (11.7)
  Dryness - Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Dryness - Non Study eye - Day 22±2 | -7.2 (15.9) | -3.6 (3.3) | -4.4 (8.8)
  Foreign body sensation - Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 1 (15 min) | -10.9 (20.0) | -28.1 (19.2) | -19.8 (11.9)
  Foreign body sensation - Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 1 (30 min) | -8.2 (20.7) | -24.0 (24.3) | -18.2 (9.6)
  Foreign body sensation - Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 15±2 (pre-dose) | -12.7 (15.3) | -15.3 (20.7) | -10.7 (9.9)
  Foreign body sensation - Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 15±2 (15 min) | -16.9 (17.9) | -27.8 (24.0) | -19.2 (11.2)
  Foreign body sensation - Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 15±2 (30 min) | -16.7 (17.6) | -23.7 (24.1) | -16.7 (9.6)
  Foreign body sensation - Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Study eye - Day 22±2 | -5.5 (12.8) | -6.1 (8.6) | -1.4 (5.9)
  Foreign body sensation - Non Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 1 (15 min) | -16.1 (12.6) | -19.1 (19.6) | -22.1 (15.7)
  Foreign body sensation - Non Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 1 (30 min) | -12.5 (13.0) | -20.6 (25.2) | -18.9 (15.1)
  Foreign body sensation - Non Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 15±2 (pre-dose) | -5.6 (21.6) | -8.2 (17.9) | -11.0 (15.1)
  Foreign body sensation - Non Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 15±2 (15 min) | -8.8 (35.4) | -16.8 (26.7) | -20.7 (17.1)
  Foreign body sensation - Non Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 15±2 (30 min) | -6.0 (33.6) | -15.7 (27.1) | -18.6 (16.7)
  Foreign body sensation - Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Foreign body sensation - Non Study eye - Day 22±2 | -1.2 (21.1) | -5.1 (4.5) | -2.1 (6.8)
  Burning/Stinging - Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 1 (15 min) | -11.7 (10.6) | -23.1 (17.2) | -18.9 (14.1)
  Burning/Stinging - Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 1 (30 min) | -10.9 (11.3) | -20.4 (18.5) | -19.0 (15.9)
  Burning/Stinging - Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 15±2 (pre-dose) | -15.5 (18.2) | -14.4 (14.0) | -6.3 (11.9)
  Burning/Stinging - Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 15±2 (15 min) | -18.3 (17.2) | -28.4 (17.5) | -18.7 (12.8)
  Burning/Stinging - Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 15±2 (30 min) | -16.0 (16.7) | -27.1 (18.2) | -13.8 (8.9)
  Burning/Stinging - Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Study eye - Day 22±2 | -10.9 (17.4) | -9.1 (9.3) | -3.3 (5.2)
  Burning/Stinging - Non Study eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 1 (15 min) | -18.9 (14.0) | -17.5 (20.1) | -19.2 (9.4)
  Burning/Stinging - Non Study eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 1 (30 min) | -15.4 (14.0) | -16.8 (21.3) | -6.2 (8.9)
  Burning/Stinging - Non Study eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 15±2 (pre-dose) | -12.1 (20.6) | -9.7 (14.2) | -6.2 (8.9)
  Burning/Stinging - Non Study eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 15±2 (15 min) | -18.6 (17.3) | -18.3 (21.5) | -15.8 (9.8)
  Burning/Stinging - Non Study eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 15±2 (30 min) | -13.2 (15.3) | -16.1 (23.4) | -13.1 (9.3)
  Burning/Stinging - Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Burning/Stinging - Non Study eye - Day 22±2 | -9.4 (21.3) | -4.8 (7.9) | -0.2 (4.7)
  Itching - Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 1 (15 min) | -9.0 (13.7) | -8.9 (11.8) | -13.0 (14.2)
  Itching - Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 1 (30 min) | -9.2 (17.4) | -8.3 (11.5) | -10.9 (12.8)
  Itching - Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 15±2 (pre-dose) | -8.1 (18.8) | -3.7 (7.1) | -6.6 (6.3)
  Itching - Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 15±2 (15 min) | -14.0 (20.1) | -7.2 (10.4) | -13.1 (13.0)
  Itching - Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 15±2 (30 min) | -11.5 (18.8) | -6.9 (10.6) | -7.7 (8.7)
  Itching - Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Itching - Study Eye - Day 22±2 | -7.2 (20.6) | -2.2 (6.0) | -3.4 (7.8)
  Itching - Non Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 1 (15 min) | -7.9 (11.8) | -8.3 (11.0) | -13.6 (9.6)
  Itching - Non Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 1 (30 min) | -7.5 (13.2) | -8.2 (11.5) | -10.4 (9.8)
  Itching - Non Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 15±2 (pre-dose) | -2.8 (14.3) | -4.8 (9.9) | -4.3 (3.8)
  Itching - Non Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 15±2 (15 min) | -7.0 (14.3) | -7.7 (11.6) | -9.1 (7.5)
  Itching - Non Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 15±2 (30 min) | -8.1 (14.8) | -7.2 (10.4) | -9.1 (9.3)
  Itching - Non Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Itching - Non Study Eye - Day 22±2 | -3.5 (16.4) | -2.1 (3.1) | -3.4 (7.4)
  Pain - Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 1 (15 min) | -10.5 (8.6) | -11.6 (15.2) | -11.9 (7.3)
  Pain - Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 1 (30 min) | -8.9 (6.4) | -10.1 (15.5) | -11.0 (10.2)
  Pain - Study Eye - Day 15 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 15 (pre-dose) | -13.7 (12.6) | -7.1 (12.9) | -5.4 (3.8)
  Pain - Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 15±2 (15 min) | -15.9 (12.1) | -11.9 (17.2) | -11.0 (6.6)
  Pain - Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 15±2 (30 min) | -14.3 (13.1) | -14.2 (17.8) | -9.4 (7.7)
  Pain - Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Pain - Study Eye - Day 22±2 | -8.3 (13.8) | -5.2 (11.8) | -0.6 (7.9)
  Pain - Non Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 1 (15 min) | -11.1 (13.3) | -4.9 (6.7) | -10.0 (8.3)
  Pain - Non Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 1 (30 min) | -10.2 (13.8) | -4.0 (9.1) | -10.0 (9.7)
  Pain - Non Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 15±2 (pre-dose) | -4.6 (9.0) | -3.8 (11.6) | -3.8 (3.9)
  Pain - Non Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 15±2 (15 min) | -7.8 (8.7) | -7.1 (12.0) | -9.7 (7.1)
  Pain - Non Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 15±2 (30 min) | -6.5 (8.8) | -7.0 (11.7) | -8.2 (7.1)
  Pain - Non Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Pain - Non Study Eye - Day 22±2 | -4.4 (9.7) | -2.1 (9.3) | 0.9 (7.3)
  Sticky feeling - Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 1 (15 min) | -7.3 (18.4) | -21.4 (16.3) | -18.7 (13.3)
  Sticky feeling - Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 1 (30 min) | -7.7 (18.6) | -22.3 (18.2) | -16.1 (10.7)
  Sticky feeling - Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 15±2 (pre-dose) | -12.6 (13.7) | -15.2 (24.4) | -9.6 (9.9)
  Sticky feeling - Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 15±2 (15 min) | -14.6 (13.0) | -24.4 (27.2) | -17.4 (12.9)
  Sticky feeling - Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 15±2 (30 min) | -12.8 (13.1) | -25.3 (24.8) | -14.8 (11.2)
  Sticky feeling - Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Study Eye - Day 22±2 | -8.7 (12.0) | -5.7 (8.8) | -1.0 (7.0)
  Sticky feeling - Non Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 1 (15 min) | -14.0 (12.1) | -15.5 (13.8) | -19.9 (13.3)
  Sticky feeling - Non Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 1 (30 min) | -12.8 (12.0) | -16.3 (16.5) | -18.1 (12.4)
  Sticky feeling - Non Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 15±2 (pre-dose) | -5.8 (9.8) | -12.4 (20.8) | -10.2 (10.4)
  Sticky feeling - Non Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 15±2 (15 min) | -4.6 (16.5) | -19.9 (23.8) | -18.9 (13.2)
  Sticky feeling - Non Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 15±2 (30 min) | -5.7 (11.7) | -18.1 (20.6) | -16.0 (12.1)
  Sticky feeling - Non Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Sticky feeling - Non Study Eye - Day 22±2 | -5.0 (10.7) | -3.7 (6.5) | -2.1 (5.9)
  Blurred vision - Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 1 (15 min) | -8.0 (9.7) | -14.2 (20.2) | -11.0 (12.3)
  Blurred vision - Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 1 (30 min) | -6.3 (9.0) | -14.9 (22.4) | -8.8 (11.9)
  Blurred vision - Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 15±2 (pre-dose) | -6.0 (7.8) | -13.9 (24.5) | -4.1 (5.1)
  Blurred vision - Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 15±2 (15 min) | -11.6 (10.5) | -18.4 (25.5) | -8.7 (8.0)
  Blurred vision - Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 15±2 (30 min) | -10.0 (10.2) | -18.2 (25.4) | -5.2 (6.8)
  Blurred vision - Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Study Eye - Day 22±2 | -3.4 (6.2) | -5.6 (8.4) | -1.0 (7.6)
  Blurred vision - Non Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 1 (15 min) | -3.8 (6.1) | -10.7 (10.8) | -9.7 (11.1)
  Blurred vision - Non Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 1 (30 min) | -4.8 (7.2) | -10.1 (15.0) | -8.3 (10.4)
  Blurred vision - Non Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 15±2 (pre-dose) | -1.8 (4.3) | -11.9 (16.1) | -4.8 (4.0)
  Blurred vision - Non Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 15±2 (15 min) | -4.8 (6.4) | -15.8 (19.9) | -8.6 (6.5)
  Blurred vision - Non Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 15±2 (30 min) | -4.2 (7.0) | -14.3 (20.8) | -5.0 (6.0)
  Blurred vision - Non Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Blurred vision - Non Study Eye - Day 22±2 | -0.7 (6.1) | -3.6 (4.9) | -1.3 (6.8)
  Photophobia - Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 1 (15 min) | -16.5 (16.2) | -23.4 (24.3) | -24.2 (14.6)
  Photophobia - Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 1 (30 min) | -14.8 (14.7) | -21.5 (27.0) | -23.2 (12.6)
  Photophobia - Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 15±2 (pre-dose) | -11.6 (16.3) | -15.6 (29.5) | -13.3 (10.6)
  Photophobia - Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 15±2 (15 min) | -18.3 (15.2) | -25.4 (31.0) | -23.7 (12.5)
  Photophobia - Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 15±2 (30 min) | -16.4 (15.5) | -25.7 (30.0) | -17.8 (9.7)
  Photophobia - Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Study Eye - Day 22±2 | -3.3 (6.5) | -6.2 (10.7) | -7.0 (13.3)
  Photophobia - Non Study Eye - Day 1 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 1 (15 min) | -13.4 (11.8) | -20.7 (24.8) | -18.7 (16.1)
  Photophobia - Non Study Eye - Day 1 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 1 (30 min) | -12.2 (10.4) | -20.0 (27.1) | -16.4 (13.3)
  Photophobia - Non Study Eye - Day 15±2 (pre-dose): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 15±2 (pre-dose) | -2.5 (6.3) | -14.2 (29.2) | -14.4 (9.4)
  Photophobia - Non Study Eye - Day 15±2 (15 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 15±2 (15 min) | -11.6 (10.3) | -16.7 (31.3) | -18.2 (13.5)
  Photophobia - Non Study Eye - Day 15±2 (30 min): number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 15±2 (30 min) | -9.8 (10.5) | -16.3 (29.3) | -15.8 (10.4)
  Photophobia - Non Study Eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Photophobia - Non Study Eye - Day 22±2 | -0.5 (5.8) | -4.8 (10.2) | -5.4 (11.8)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Dryness - Study eye - Day 15±2 The model included fixed effect terms for time point, baseline covariate (i.e. the day 1 - pre-dose value) and treatment. Time point was specified as a repeated measurement; Test type: Superiority; p = 0.3474, ANOVA; Analysis of variance for repeated measures; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-3.3 to 9.1]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Dryness - Study eye - Day 15±2; Test type: Superiority; p = 0.1327, ANOVA; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-8.2 to 4.3]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Dryness - Study eye - Day 15±2; Test type: Superiority; p = 0.1327, ANOVA; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-11.2 to 1.6]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Foreign body sensation - Study eye - Day 15±2; Test type: Superiority; p = 0.2237, ANOVA; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-2.5 to 10.0]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Foreign body sensation - Study eye - Day 15±2; Test type: Superiority; p = 0.4905, ANOVA; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-8.4 to 4.1]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Foreign body sensation - Study eye - Day 15±2; Test type: Superiority; p = 0.0687, ANOVA; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-12.3 to 0.5]
Statistical Analysis 7: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Study eye - Day 15±2; Test type: Superiority; p = 0.7609, ANOVA; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-4.2 to 5.6]
Statistical Analysis 8: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Study eye - Day 15±2; Test type: Superiority; p = 0.6428, ANOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-6.0 to 3.8]
Statistical Analysis 9: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Study eye - Day 15±2; Test type: Superiority; p = 0.4599, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-6.9 to 3.2]
Statistical Analysis 10: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Study eye - Day 15±2; Test type: Superiority; p = 0.4217, ANOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-4.6 to 10.5]
Statistical Analysis 11: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Study eye - Day 15±2; Test type: Superiority; p = -2.5, ANOVA; Mean Difference (Final Values) = 0.5030, 95% CI 2-sided [-10.0 to 5.0]
Statistical Analysis 12: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Study eye - Day 15±2; Test type: Superiority; p = 0.4599, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-6.9 to 3.2]
Statistical Analysis 13: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Study eye - Day 15±2; Test type: Superiority; p = 0.6157, ANOVA; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.6 to 4.4]
Statistical Analysis 14: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Study eye - Day 15±2; Test type: Superiority; p = 0.9120, ANOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-3.7 to 3.3]
Statistical Analysis 15: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Study eye - Day 15±2; Test type: Superiority; p = 0.5463, ANOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.6 to 2.5]
Statistical Analysis 16: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky Feeling - Study eye - Day 15±2; Test type: Superiority; p = 0.9065, ANOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-5.9 to 5.3]
Statistical Analysis 17: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky Feeling - Study eye - Day 15±2; Test type: Superiority; p = 0.5065, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.3 to 3.7]
Statistical Analysis 18: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky Feeling - Study eye - Day 15±2; Test type: Superiority; p = 0.5977, ANOVA; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-7.1 to 4.2]
Statistical Analysis 19: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred Vision - Study eye - Day 15±2; Test type: Superiority; p = 0.2785, ANOVA; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-6.3 to 1.9]
Statistical Analysis 20: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred vision - Study eye - Day 15±2; Test type: Superiority; p = 0.7454, ANOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.6 to 3.3]
Statistical Analysis 21: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred vision - Study eye - Day 15±2; Test type: Superiority; p = 0.4588, ANOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-2.7 to 5.9]
Statistical Analysis 22: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Study eye - Day 15±2; Test type: Superiority; p = 0.2812, ANOVA; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-3.7 to 12.3]
Statistical Analysis 23: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Study eye - Day 15±2; Test type: Superiority; p = 0.6811, ANOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-6.5 to 9.8]
Statistical Analysis 24: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Study eye - Day 15±2; Test type: Superiority; p = 0.5169, ANOVA; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-10.8 to 5.6]
Statistical Analysis 25: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Dryness - Non Study eye - Day 15±2; Test type: Superiority; p = 0.7874, ANOVA; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-5.9 to 7.8]
Statistical Analysis 26: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Dryness - Non Study eye - Day 15±2; Test type: Superiority; p = 0.8299, ANOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-7.6 to 6.1]
Statistical Analysis 27: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Dryness - Non Study eye - Day 15±2; Test type: Superiority; p = 0.6386, ANOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-8.7 to 5.4]
Statistical Analysis 28: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Foreign body sensation - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0132, ANOVA; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [1.3 to 10.2]
Statistical Analysis 29: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 1, analysis 28]; Test type: Superiority; p = 0.7177, ANOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.3 to 3.7]
Statistical Analysis 30: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 1, analysis 28]; Test type: Superiority; p = 0.0077, ANOVA; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-11.2 to -1.9]
Statistical Analysis 31: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0301, ANOVA; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [0.6 to 10.0]
Statistical Analysis 32: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Non Study eye - Day 15±2; Test type: Superiority; p = 0.8657, ANOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-4.3 to 5.1]
Statistical Analysis 33: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Burning/Stinging - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0440, ANOVA; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-9.7 to -0.1]
Statistical Analysis 34: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Non Study eye - Day 15±2; Test type: Superiority; p = 0.1351, ANOVA; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-1.4 to 9.6]
Statistical Analysis 35: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Non Study eye - Day 15±2; Test type: Superiority; p = 0.8821, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-6.0 to 5.2]
Statistical Analysis 36: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Itching - Non Study eye - Day 15±2; Test type: Superiority; p = 0.1208, ANOVA; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-10.3 to 1.3]
Statistical Analysis 37: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Non Study eye - Day 15±2; Test type: Superiority; p = 0.9440, ANOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.3 to 3.5]
Statistical Analysis 38: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Non Study eye - Day 15±2; Test type: Superiority; p = 0.4903, ANOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-2.2 to 4.5]
Statistical Analysis 39: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Pain - Non Study eye - Day 15±2; Test type: Superiority; p = 0.5364, ANOVA; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.3 to 4.3]
Statistical Analysis 40: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky feeling - Non Study eye - Day 15±2; Test type: Superiority; p = 0.5100, ANOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-2.9 to 5.7]
Statistical Analysis 41: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky feeling - Non Study eye - Day 15±2; Test type: Superiority; p = 0.1132, ANOVA; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-0.9 to 7.8]
Statistical Analysis 42: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Sticky feeling - Non Study eye - Day 15±2; Test type: Superiority; p = 0.3457, ANOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-2.4 to 6.5]
Statistical Analysis 43: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred vision - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0185, ANOVA; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [0.8 to 7.9]
Statistical Analysis 44: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred vision - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0408, ANOVA; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [0.2 to 7.1]
Statistical Analysis 45: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Blurred vision - Non Study eye - Day 15±2; Test type: Superiority; p = 0.6992, ANOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-4.4 to 3.0]
Statistical Analysis 46: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Non Study eye - Day 15±2; Test type: Superiority; p = 0.0905, ANOVA; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-1.0 to 12.8]
Statistical Analysis 47: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Non Study eye - Day 15±2; Test type: Superiority; p = 0.3054, ANOVA; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-3.4 to 10.4]
Statistical Analysis 48: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Analysis of variance on changes from baseline in ocular tolerability - Photophobia - Non Study eye - Day 15±2; Test type: Superiority; p = 0.5024, ANOVA; Mean Difference (Final Values) = 0.5024, 95% CI 2-sided [-9.6 to 4.8]

2. Primary Outcome: Treatment-emergent Adverse Events (TEAEs) Assessed Throughout the Study
Description: TEAEs included all AEs occurring or worsening after the first dose of IMD. These comprise AEs during the treatment and follow-up period. For TEAE, the number of events was provided.
  At each visit (Visit 1 which took place at Day 1; Visit 2 which took place at day 15 ± 2; Visit 3, i.e. final visi FU, at Day 22 ± 2/ETV), patients could spontaneously report any physical or medical occurrence and the investigator or designee inquired about the occurrence of TEAEs by asking specific questions. Any untoward (unfavorable & unintended) change in subject's medical conditions was to be reported as an AE. Changes in any protocol-specific ocular or systemic parameter evaluated during the study were to be reviewed by the investigator. In addition, each patient's response to any questionnaire was to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in a protocol-specific parameter or questionnaire response clinically relevant was to be reported as an AE.
Time Frame: From baseline (Day 1 - pre-dose) to day 22±2
Population: The Safety population (SAF) included all patients who received and used at least once the IMDs (Lubricin or Vismed ®).
Measure: Number; unit: events
Groups:
- Lubricin 20µg/ml (SAF): Lubricin 20µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 20µg/ml: Lubricin 20µg/ml eye drops
- Lubricin 50µg/ml (SAF): Lubricin 50µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 50µg/ml: Lubricin 50µg/ml eye drops
- Sodium Hyaluronate 0.18% (SAF): Vismed® 0.18% Sodium hyaluronate (HA) eye drops
  Comparator was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2.
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Sodium hyaluronate 0.18%: Sodium hyaluronate (HA) 0.18% eye drops
Arm/Group | Lubricin 20µg/ml (SAF) | Lubricin 50µg/ml (SAF) | Sodium Hyaluronate 0.18% (SAF)
Number analyzed (Participants) | 10 | 10 | 10
events | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Ocular Surface Vital Staining With Fluorescein (Oxford Scale)
Description: The corneal fluorescein staining was graded by using the Oxford scheme to assess cornea and conjunctiva epithelium damage. It was performed after instillation of sodium fluoresce into the inferior conjunctival cul-de-sac of each eye with the aid of a slit lamp at 10X magnification using cobalt blue illumination.
  The Oxford scale grading divides corneal staining into six groups for each panel, based on the severity [from 0 (absent) to 5 (severe)]. The corneal staining is represented by punctate dots on a series of panels (panel A=grade 0 to panel >E=grade 5). Staining ranges from 0-5 for each panel, and 0-15 for the total exposed inter-palpebral conjunctiva and cornea.
  The examiner selected the appropriate grade that best represented the state of corneal staining intuitional. The higher the grade, the worst is the overall outcome value.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: The Full Analysis Set (FAS) population included all randomised patients, who received and used at least once the investigational device (Lubricin or Vismed®). Please note that for participants, study eye and non-study eye values were assessed and reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
score on a scale
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 15±2 | -0.3 (0.5) | -0.7 (0.5) | -0.6 (0.5)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 22±2 | -0.3 (0.5) | -0.6 (0.5) | -0.2 (0.4)
  Non Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 15±2 | -0.3 (0.5) | -0.3 (0.5) | 0 (0)
  Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 22±2 | -0.1 (0.3) | -0.1 (0.3) | 0 (0)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1226, Student t-test pooled; Student t-test with pool method for estimating common variance on changes from baseline in ocular surface vital staining; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.2854, Student t-test pooled; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in ocular surface vital staining - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.6525, Student t-test pooled; Student t-test pooled method for estimating common variance on changes from baseline in ocular surface vital staining -; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.4]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.8843, Student t-test pooled; Student t-test pooled method for estimating common variance on changes from baseline in ocular surface vital staining -; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.0806, Student t-test pooled; Student t-test pooled method for estimating common variance on changes from baseline in ocular surface vital staining; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.0]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.0628, Student t-test pooled; Student t-test pooled method for estimating common variance on changes from baseline in ocular surface vital staining; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.0]

4. Secondary Outcome: Change From Baseline in Schirmer-I Test (Without Anaesthesia)
Description: The Schirmer test Type I (without anaesthesia) was performed to measure aqueous tear secretion prior to the instillation of any dilating or anaesthetic eye drops. The rounded bent end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schirmer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). The longer the wetted length, the healthier the status of the eye.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/5min
Units Other Than Participants: eyes
Groups:
- Lubricin 20µg/ml (FAS): Lubricin 20µg/ml eye drops solution
  Test investigational device was instilled t.i.d. (three times a day) approximately every 6 h, from day 1 to day 15±2. Test investigational device was instilled
  All the patients instilled their assigned IMD into both eyes, unless only one eye met the eligibility criteria. If just one eye met the eligibility criteria, that was identified as the "Study/Primary eye". If both eyes met the eligibility criteria, the worst one (highest VAS average score) was chosen as "Study/Primary eye". In the event that the mean VAS score was equal in both eyes, right eye was to be chosen as "Study/Primary eye".
  The investigator instilled the morning study dose on Day 1 then the patients self-instilled the drops at home/site, as applicable.
  After the end of the treatment period, all the subjects could use any ocular topical treatment allowed, including other artificial tears/lubricants as prescribed by the treating physician, from day 15±2 to day 21±2.
  Lubricin 20µg/ml: Lubricin 20µg/ml eye drops
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
mm/5min
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 15±2 | 0.7 (0.5) | 0.3 (0.7) | 0.6 (0.5)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 22±2 | 0.4 (1.0) | 0.1 (0.8) | 0.2 (1.6)
  Non Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 15±2 | 0.4 (0.5) | -0.2 (1.1) | -0.1 (0.6)
  Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 22±2 | 0.0 (0.7) | -0.7 (0.7) | -0.2 (1.1)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in Schirmer-I test - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.2004, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in Schirmer-I test - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.5413, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in Schirmer-I test - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4607, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in Schirmer-I test - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1248, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.2 to 1.4]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in Schirmer-I test - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.0624, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.0 to 1.1]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in Schirmer-I test - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.7927, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.8]

5. Secondary Outcome: Change From Baseline in Permanence of Lubricin on the Ocular Surface - Tear Film Break-up Time (TFBUT)
Description: TFBUT was measured by determining the time to tear break-up. The TFBUT test was performed after instillation of 5 μl of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner monitored the integrity of the tear film, noting the time it took to form lacunae (clear spaces in the tear film) from the time that the eye was opened after the last blink. This measurement was performed within 10 seconds maximum. The TFBUT was measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differed by more than 2 seconds, a third reading was taken. The TFBUT value was the average of the 2 or 3 measurements. Generally, a TFBUT value of 10-35 seconds was considered normal. A value of less than 10 seconds was usually suspicious and may indicate tear film instability. The higher the value, the better the outcome.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
seconds
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 15±2 | 0.9 (0.7) | 0.9 (0.6) | 0.8 (0.8)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 22±2 | 0.9 (0.9) | 0.9 (0.6) | 0.4 (0.7)
  Non Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 15±2 | 0.2 (0.8) | 0.6 (0.7) | 0.0 (0.7)
  Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 22±2 | 0.2 (0.8) | 0.4 (1.7) | -0.2 (0.7)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in TFBUT - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.9717, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.7]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.7386, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.9]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in TFBUT - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.7498, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.8]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in TFBUT - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.3229, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.4]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in TFBUT - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.5700, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.5 to 0.9]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in TFBUT - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1197, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.2 to 1.3]

6. Secondary Outcome: Change From Baseline in Best Corrected Distance Visual Acuity (BCDVA) - ETDRS Score
Description: Best corrected visual acuity (BCDVA) was determined by careful refraction according to the standard protocol for refraction. Chart 1 was used for testing the VA of the right eye; Chart 2 for the left eye; and Chart R for refraction only. Retroilluminated standard Early Treatment of Diabetic Retinopathy Study (ETDRS) charts were used. They had 5 Sloan letters on each line of equal difficulty, and there was a geometric progression in letter size from line to line. VAS awarded one point for every letter correctly guessed. A distance of 4 meters was required between the subject's eyes and the VA chart. When a subject cannot read at least 20 letters on the chart at 4 meters, the subject was tested at 1 meter. If 20 or more letters were read at 4 meters, the VAS for that eye was recorded as the number of letters correct at 4 meters plus 30. Otherwise, the VAS was the number of letters read correctly at 1 meter plus the number read at 4 meters. The higher the score the better the outcome.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
score on a scale
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 15±2 | 0.4 (0.7) | 0.4 (0.5) | 0.3 (0.5)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 22±2 | 0.1 (0.6) | 0.4 (1.5) | 0.0 (1.7)
  Non Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 15±2 | -0.1 (0.9) | 0.2 (0.4) | -0.1 (0.6)
  Non Study eye - day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - day 22±2 | -0.1 (0.6) | 0.1 (0.6) | -0.2 (0.7)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in BCDVA - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.8787, Student t-test pooled; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in BCDVA - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.8159, Student t-test pooled; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in BCDVA - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.6525, Student t-test pooled; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in BCDVA - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.3340, Student t-test pooled; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in BCDVA - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.9749, Student t-test pooled; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in BCDVA - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1984, Student t-test pooled; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.2 to 0.9]

7. Secondary Outcome: Change From Baseline in SANDE (Symptom Assessment in Dry Eye) Questionnaire Scores
Description: The SANDE (Symptom Assessment in Dry Eye) questionnaire was a short questionnaire to evaluate both dry eye frequency and severity by using a 100 mm VAS. The subject symptoms of ocular dryness and/or irritation were quantified on the scale based on two questions that assess both severity and frequency of symptoms. For the assessment, the subjects marked on the 100 mm VAS line the point that they felt represented their perception of their current state. The VAS score was determined by measuring in millimeters from the left hand end of the line to the point that the subject marked. The SANDE scores was then evaluated for the 2 questions severity (0-100) and frequency (0-100), where 0 was the best condition and 100 marked the worst condition.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: The Full Analysis Set (FAS) population included all randomised patients, who received and used at least once the investigational device (Lubricin or Vismed®).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
mm
  Frequency of Symptoms - Day 15±2 | -14.6 (12.9) | -17.6 (15.0) | -7.7 (4.4)
  Frequency of Symptoms - Day 22±2 | -11.9 (9.8) | -11.9 (7.4) | -2.7 (6.9)
  Severity of Symptoms - Day 15±2 | -11.2 (11.2) | -15.0 (12.9) | -7.1 (4.5)
  Severity of Symptoms - Day 22±2 | -7.4 (10.7) | -7.2 (10.5) | -2.7 (4.1)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in SANDE scores - Frequency of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.6497, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-10.5 to 16.4]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in SANDE scores - Frequency of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.1443, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-16.5 to 2.6]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in SANDE scores - Frequency of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.0751, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-20.9 to 1.1]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in SANDE scores - Severity of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.5015, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-7.9 to 15.5]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in SANDE scores - Severity of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.3217, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-12.5 to 4.4]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in SANDE scores - Severity of symptoms - Day 15±2 pre-dose; Test type: Superiority; p = 0.1026, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-17.5 to 1.8]

8. Secondary Outcome: Change From Baseline in Slit Lamp Examination (SLE) Values
Description: The Slit Lamp Examination was used to examine the structures of the eye (eyelids, lashes, conjunctiva, cornea, lens, iris and anterior chamber) according to different scales: Eyelid - Meibomian glands (from 0-none to 3-severe), Eyelid - Erythema (from 0-none to 4-very severe), Eyelid - Oedema (from 0-none to 4-very severe), Lashes (0-normal 1-abnormal), Conjunctiva - Erythema (from 0-none to 3-severe), Conjunctiva - Oedema (from 0-none to 4-very severe), Lens (to 0-no opacification to 3-severe opacification), Iris (0-normal 1-abnormal), Anterior chamber inflammation (from 0-none to 3-severe), Cornea transparency (from 0-completely transparent to 4-complete cornea opacity), Cornea neovascularization (0-absence of vascularization to 4- neovascularization between 270° and 360°). The higher the score the worse the outcome. There was not a total score.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
score on a scale
  Eyelid - Meibomian glands (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid - Meibomian glands (Study eye) - Day 15±2 | -0.1 (0.3) | -0.1 (0.3) | -0.1 (0.3)
  Eyelid - Meibomian glands ( Non Study eye) - Day15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid - Meibomian glands ( Non Study eye) - Day15±2 | -0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid - Meibomian glands (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid - Meibomian glands (Study eye) - Day 22±2 | -0.1 (0.3) | -0.1 (0.3) | -0.2 (0.4)
  Eyelid - Meibomian glands (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid - Meibomian glands (Non Study eye) - Day 22±2 | -0.1 (0.3) | -0.1 (0.3) | -0.1 (0.3)
  Eyelid erythema (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid erythema (Study eye) - Day 15±2 | -0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid erythema (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid erythema (Non Study eye) - Day 15±2 | -0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid erythema (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid erythema (Study eye) - Day 22±2 | -0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid erythema (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid erythema (Non Study eye) - Day 22±2 | -0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid Oedema (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid Oedema (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid Oedema (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid Oedema (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid Oedema (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid Oedema (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Eyelid Oedema (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Eyelid Oedema (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Lashes (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Lashes (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Lashes (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Lashes (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - erythema (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - erythema (Study eye) - Day 15±2 | -0.1 (0.3) | -0.2 (0.4) | -0.3 (0.5)
  Conjunctiva - erythema (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - erythema (Non Study eye) - Day 15±2 | -0.1 (0.3) | -0.4 (0.5) | 0.1 (0.3)
  Conjunctiva - erythema (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - erythema (Study eye) - Day 22±2 | -0.1 (0.3) | 0.0 (0.5) | 0.1 (0.6)
  Conjunctiva - erythema (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - erythema (Non Study eye) - Day 22±2 | -0.1 (0.3) | -0.1 (0.3) | 0.2 (0.4)
  Conjunctiva - oedema (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - oedema (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - oedema (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - oedema (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - oedema (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - oedema (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - oedema (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Conjunctiva - oedema (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lens (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Lens (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lens (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Lens (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lens (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Lens (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Lens (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Lens (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Iris (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Iris (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Iris (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 20 | 9
  Iris (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Iris (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Iris (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Iris (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Iris (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Anterior chamber inflammation (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Anterior chamber inflammation (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Anterior chamber inflammation (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Anterior chamber inflammation (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea transparency (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea transparency (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea transparency (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea transparency (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea neovascularization (Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Non Study eye) - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea neovascularization (Non Study eye) - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea neovascularization (Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Non Study eye) - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Cornea neovascularization (Non Study eye) - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Meibomian Glands - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Meibomian Glands - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Erythema - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Erythema - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.4101, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Oedema - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Eyelid - Oedema - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 16]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 16]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lashes - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Conjunctiva - Erythema - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.5267, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 25]; Test type: Superiority; p = 0.2633, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 25]; Test type: Superiority; p = 0.6552, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Conjunctiva - Erythema - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1262, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 28]; Test type: Superiority; p = 0.2094, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 28]; Test type: Superiority; p = 0.0377, Wilcoxon (Mann-Whitney); Hodges Lehmann estimation = -1.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 31: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Conjunctiva - Oedema - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 32: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 31]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 33: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 31]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 34: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Conjunctiva - Oedema - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 35: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 34]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 36: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 34]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 37: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 38: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 39: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 40: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 41: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 42: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Lens - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 43: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 44: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 45: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 46: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 47: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 48: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Iris - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 49: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Anterior chamber inflammation - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 50: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 49]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 51: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 49]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 52: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Anterior chamber inflammation - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 53: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 52]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 54: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 52]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 55: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Cornea transparency - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 56: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 55]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 57: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 55]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 58: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Cornea transparency - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 59: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 58]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 60: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 58]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 61: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Cornea neovascularization - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 62: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 61]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 63: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 61]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 64: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Wilcoxon Rank Sum Test on changes from baseline in SLE examination scores - Cornea neovascularization - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 65: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 64]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 66: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); [analysis description as in outcome 8, analysis 64]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in IOP (Intraocular Pressure)
Description: The IOP (intraocular pressure) of the eye was determined by the balance between the amount of aqueous humor that the eye marked and ease with which it leaved the eye. IOP was performed using Goldmann applanation tonometry after the instillation of a topical anaesthetic. The Goldmann applanation tonometer measured the force necessary to flatten a corneal area of 3.06 mm diameter. At this diameter, the resistance of the cornea to flattening was counterbalanced by the capillary attraction of the tear film meniscus for the tonometer head. The IOP (in mm Hg) equals the flattening force (in grams) multiplied by 10. IOP was measured in both eyes after completion of all SLEs to avoid potential interference with the other evaluations. Both eyes were tested. Normal eye pressure was between 10 to 21 mmHg. High ocular pressure was greater than 21 mmHg.
Time Frame: Day 15±2 (Visit 2); Day 22±2 (Visit 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
mmHg
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 15±2 | 0.2 (1.9) | -0.3 (2.3) | 0.8 (1.4)
  Non study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 9
  Non study eye - Day 15±2 | 0.1 (0.7) | 0.6 (2.0) | 0.7 (1.7)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Study eye - Day 22±2 | -0.5 (2.0) | -0.6 (2.6) | -1.7 (3.9)
  Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 9
  Non Study eye - Day 22±2 | -0.9 (1.6) | 1.4 (3.0) | -1.3 (1.8)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in IOP - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.5842, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.6]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in IOP - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4606, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.2 to 1.0]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in IOP - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.2319, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.0 to 0.8]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in IOP - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.6018, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.3 to 1.4]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in IOP - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.4857, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.2 to 1.1]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in IOP - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.9015, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.0 to 1.8]

10. Secondary Outcome: Change From Baseline in Corneal Sensitivity by Cochet-Bonnet Aesthesiometry
Description: The Cochet-Bonnet aesthesiometer contained a thin, retractable, nylon monofilament that extended up to 6 cm in length. Variable pressure could be applied to the cornea by adjusting the monofilament length. The monofilament length ranged from 6 to 0.5 cm. As the monofilament length was decreased the pressure increased from 11 mm/gm to 200 mm/gm. Corneal sensation was measured in the affected eye(s) in the central area of the cornea using a Cochet Bonnet aesthesiometer before the instillation of any dilating or anesthetic eye drops. The length of the filament in cm at which the patient corneal sensation was observed for the tested area of the cornea was reported. With decreasing length of monofilament, the corneal touch threshold increased and the corneal sensitivity decreased. Therefore, decreasing the length of monofilament was proportional to decreased corneal sensitivity.
Time Frame: From baseline (Day 1 pre-dose) to Day 15±2 and Day 22±2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: eyes
Arm/Group | Lubricin 20µg/ml (FAS) | Lubricin 50µg/ml (FAS) | Sodium Hyaluronate (FAS)
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
cm
  Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 18
  Study eye - Day 15±2 | 0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0)
  Non Study eye - Day 15±2: number analyzed (eyes) | 10 | 10 | 18
  Non Study eye - Day 15±2 | 0.0 (0.0) | 0.0 (0.0) | -0.1 (0.3)
  Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 18
  Study eye - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Non Study eye - Day 22±2: number analyzed (eyes) | 10 | 10 | 18
  Non Study eye - Day 22±2 | 0.0 (0.0) | 0.0 (0.0) | -0.2 (0.4)
Statistical Analysis 1: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in corneal sensitivity - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.3574, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 2: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in corneal sensitivity - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.3574, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 3: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in corneal sensitivity - Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 00, Student t-test pooled — P-value is NA due to the measured values of corneal sensitivity equal to zero; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 4: Comparison: Lubricin 20µg/ml (FAS) vs Lubricin 50µg/ml (FAS); Student t-test on changes from baseline in corneal sensitivity - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 00, Student t-test pooled — P-value is NA due to the measured values of corneal sensitivity equal to zero; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 5: Comparison: Lubricin 20µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in corneal sensitivity - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 6: Comparison: Lubricin 50µg/ml (FAS) vs Sodium Hyaluronate (FAS); Student t-test on changes from baseline in corneal sensitivity - Non Study eye - Day 15±2 pre-dose; Test type: Superiority; p = 0.1, Student t-test pooled; Pooled method for estimating common variance was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse events data were collected was from Day 1 (Visit 1) to Day 22±2 (Final Visit - Follow up) or Early Termination Visit (ETV).
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medical product and which did non necessarily have a causal relationship with this treatment. AE = any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
  No TEAE occurred during the study, neither serious, nor non serious.
Arm/Group | Lubricin 20µg/ml (SAF) | Lubricin 50µg/ml (SAF) | Sodium Hyaluronate 0.18% (SAF)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03031327/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03031327/SAP_001.pdf